CLINICAL TRIAL: NCT01088009
Title: A Prospective, Randomised, Open-label, Multi-centre Study to Compare Three Chronic Hepatitis B (CHB) Treatment Strategies Over a 2year Period in Chinese HBeAg Positive CHB Patients
Brief Title: Efficacy Optimizing Research of Lamivudine Therapy
Acronym: EXPLORE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Major Science and Technology Special Project of China Eleventh Five-year (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOH-02
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-09

CONDITIONS: Compensated Chronic Hepatitis B
Keywords: chronic hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Lamivudine; adefovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- early add-on (Experimental)
  Interventions: Drug: lamivudine
- SOC (Active Comparator): Patients will receive oral lamivudine 100mg,daily for 104 weeks, if HBV DNA breakthrough, add on oral adefovir 10mg daily
  Interventions: Drug: lamivudine
- De-novo combination (Other): patients in this arm will receive oral lamivudine 100mg and adefovir 10mg for 104 weeks
  Interventions: Drug: lamivudine, adefovir

INTERVENTIONS:
Drug: lamivudine — patients in this arm will receive oral lamivudine 100mg,daily for 24 weeks; if patients with HBV DNA higher than 1000 copies/ml at week 24, add on adefovir to week 104; otherwise, keep lamivudine monotherapy to week 104
  Arms: early add-on
Drug: lamivudine — Patients will receive oral lamivudine 100mg,daily for 104 weeks, if HBV DNA breakthrough, add on oral adefovir 10mg daily
  Arms: SOC
Drug: lamivudine, adefovir — patients in this arm will receive oral lamivudine 100mg daily and adefovir 10mg for 104 weeks
  Arms: De-novo combination

SUMMARY:
The purpose of this study is to compare the adefovir early add-on to rescue therapy strategy, and also explore the efficacy of Lamivudine and adefovir de-novo combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-65 years;
* Capable of understanding and signing the informed consent. Willing to comply with the study requirements;
* Serum HBsAg and HBeAg positive at study screening; Documented chronic hepatitis B infection determined by the presence of serum HBsAg for at least 6 months;

Exclusion Criteria:

* History of decompensated liver function, or current signs/symptoms of decompensation e.g. ascites, variceal bleeding, encephalopathy or spontaneous peritonitis;
* other protocol defined inclusion/exclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2010-03; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
the proportion of virological breakthrough with confirmed Lamivudine resistant mutants | during 104 weeks study period

SECONDARY OUTCOMES:
proportion of subjects with hepatitis B virus (HBV) DNA≤300 copies/mL | week 104
Reduction of serum HBV DNA level from baseline (log10 copies/mL) to week 104 | baseline, week 104
The proportion of subjects with ALT normalization at week 104 | week 104
The proportion of subjects with HBeAg loss and seroconversion at week 104 | week 104
The proportion of subjects with HBsAg loss and seroconversion rates at week 104 | week 104

CONTACTS AND LOCATIONS:
Overall Officials: JinLin Hou, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (24):
- China (24):
  - Beijing Ditan Hospita, Beijing, Beijing Municipality
  - Beijing Friendship Hospital Attached to the Capital Medical University, Beijing, Beijing Municipality
  - BeiJing YouAn Hospital ,Capital Medical University, Beijing, Beijing Municipality
  - Department of infectious disease, First Hospital of Peking University, Beijing, Beijing Municipality
  - People'S Hospital Under Beijnig University, Beijing, Beijing Municipality
  - The Second Affiliated of ChongQing University of Medical Science, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Department of infectious disease, Nanfang Hospital, Guangzhou, Guangdong
  - GuangDong Provincial People's hospital, Guangzhou, Guangdong
  - First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central-South Univrsity, Changsha, Hunan
  - First Hospital .Jilin Unniversity, Changchun, Jilin
  - ShengJing Hospital of China Medical University, Shenyang, Liaoning
  - JiNan Infectious Diseases Hospital, Jinan, Shandong
  - Changhai Hospital affiliated to Second Military Medical University, Shanghai, Shanghai Municipality
  - Huashan Hospital，Fudan University, Shanghai, Shanghai Municipality
  - No.85 Hospital of PLA, Shanghai, Shanghai Municipality
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - Tangdu Hospital, XiAn, Shanxi
  - West China Hospital.SiChuan University, Chengdu, Sichuan
  - HangZhou No.6 People Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of College of Medicine ，Zhejiang University, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Xiang KH, Michailidis E, Ding H, Peng YQ, Su MZ, Li Y, Liu XE, Dao Thi VL, Wu XF, Schneider WM, Rice CM, Zhuang H, Li T. Effects of amino acid substitutions in hepatitis B virus surface protein on virion secretion, antigenicity, HBsAg and viral DNA. J Hepatol. 2017 Feb;66(2):288-296. doi: 10.1016/j.jhep.2016.09.005. Epub 2016 Sep 17. PMID 27650283